CLINICAL TRIAL: NCT03375931
Title: The Effects of Preoperative Prayer on Postoperative Quality of Recovery in Patients Undergoing Thyroidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4-2017-0251
Record Dates: First submitted 2017-12-05; First posted 2017-12-18 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Thyroid Cancer
Keywords: Quality of Recovery 40 Questionaries
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Faith Healing

STUDY DESIGN:
Intervention Model Description: Prospective Randomized open study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prayer group (Experimental)
  Interventions: Behavioral: Prayer
- non-prayer group (Active Comparator)
  Interventions: Behavioral: non-prayer

INTERVENTIONS:
Behavioral: Prayer — If the patient wishes to pray, the anesthesiologist will pray for one minute before anesthesia.
  Arms: prayer group
Behavioral: non-prayer — If the patient does not want to pray, the anesthesiologist does anesthesia without praying.
  Arms: non-prayer group

SUMMARY:
physiological end-point, incidence of adverse events, and changes in psychological status.

In the past, physiological goals, major morbidity and mortality were used as indicators of recovery after surgery. However, major morbidity and mortality rates were extremely low due to the development of surgery and anesthesia techniques, and measurements of these indicators do not adequately reflect postoperative recovery. On the other hand, the measurement of the patient's health status or quality of life has become an important metric in many clinical studies. The Quality of Recovery 40 Questionnaire (QoR-40) is a multidimensional tool that specifically assesses and develops anesthetic and postoperative health conditions. Severance Hospital is conducting an anesthesiologist-led prayer for the patient only for the desired patient before anesthesia. Although it may be expected that this preoperative airway may improve the quality of recovery after anesthesia / surgery by reducing patient anxiety, there is no objective study on this. The aim of this study was to investigate the effect of preoperative preoperative airway on the quality of postoperative recovery in patients who underwent thyroidectomy for thyroid cancer. I want to see. In addition, we will investigate whether preoperative airway affects sympathetic nervous system during surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients between 20 and 70 years old under ASA 3.
* obtaining written informed consent from the patients who were undergoing thyroidectomy.
* weights under 90 kg and BMI under 30

Exclusion Criteria:

* emergency operation
* re-operation
* combined surgery over 4 departments
* cardiac disease (unstable angina, congestive heart failure, valvular heart disease)
* Ventricular conduction abnormality
* prior pacemaker insertion
* uncontrolled hypertension (diastolic blood pressure > 110mmHg)
* bradycardia (HR < 40 Bpm)
* cerebral vascular disease (cerebral hemorrhage, cerebral ischemia)
* hepatic or renal failure
* patients who take antiarrythmic agent
* neurological or psychiatric illnesses
* foreigner and patient who can not read the letter

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-12-15 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
QoR40 on POD1 | within the first 1 day after surgery
  On the first day after surgery, visit the patient and give the QoR 40 to the patient to fill out a questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No